CLINICAL TRIAL: NCT04237363
Title: Recovery of Walking Without Epidural Spinal Cord Stimulation in Adults With Complete Spinal Cord Injury
Brief Title: Recovery of Walking in Persons With Complete Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Middle Tennessee State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-310
Record Dates: First submitted 2020-01-15; First posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injury; Exercise; Walking; Aquatics
MeSH Terms: conditions — Spinal Cord Injuries; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): Walk training
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Underwater treadmill training and supplemental overground walk training

SUMMARY:
We documented the impact of 1 year of underwater treadmill training and supplemental overground walk training in five adults with chronic motor-complete SCI (cSCI) who had not undergone programmed epidural spinal cord stimulation (eSCS).

DETAILED DESCRIPTION:
Regular exposure to self-initiated treadmill walking in water, a unique sensorimotor exercise setting that makes stepping movements easier to perform, may capitalize on the adaptability of the neuromuscular system and enhance locomotor function in persons with cSCI who have not undergone eSCS. In our study, a combined aquatics- and land-based approach to gait training was employed over a 12-month period that featured underwater treadmill training and supplemental overground walk training.

ELIGIBILITY:
Inclusion Criteria

* At least 21 years of age
* Presence of traumatic or non-traumatic spinal cord injury for at least 1 year
* Medical diagnosis of paraplegia (T1 or below)

Exclusion Criteria

* Presence of complex comorbidities that could limit involvement in training activities
* Surgical implantation or removal of a medical device six months prior to training
* Skin breakdown
* Use of electrical implants to promote ambulation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-07-05 (Actual); Primary Completion 2013-08-06 (Actual); Study Completion 2013-08-06 (Actual)

PRIMARY OUTCOMES:
Overground walking capacity | Change from Baseline WISCI-II score at 6 months and 12 months
  Walking Capacity for Spinal Cord Injury (WISCI-II)

CONTACTS AND LOCATIONS:
Overall Officials: Don W Morgan, PhD, Study Director — Middle Tennessee State University; Sandra L Stevens, PhD, PT, Principal Investigator — Middle Tennessee State University